CLINICAL TRIAL: NCT02197273
Title: Efficacy of Liposomal Bupivacaine Versus Standard Analgesia in Pain Management of Total Joint Arthroplasty
Brief Title: Liposomal Bupivacaine Versus Standard Analgesia in Total Joint Arthroplasty (TJA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Deborah Napier, Clinical Outcomes Manager, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OH1-14-00529
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis, Shoulder
Keywords: Total knee arthroplasty; Total shoulder arthroplasty; Total hip arthroplasty; Total joint arthroplasty; Hip replacement; Knee replacement; Shoulder replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — Bupivacaine; Ropivacaine; Fentanyl; Methylprednisolone Hemisuccinate; Morphine; Sodium Chloride; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care analgesia (Active Comparator): Total Hip Arthroplasty (THA):
  All patients will receive a spinal anesthetic using Fentanyl and Bupivacaine
  Injection into capsular tissue after placement of the acetabular component:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  Total Knee Arthroplasty (TKA):
  All patients will receive a spinal anesthetic using Fentanyl and Bupivacaine All patients will receive an adductor canal block of 0.25% Bupivacaine w/epinephrine 30cc
  Injection into posterior capsule of the knee:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  Total Shoulder Arthroplasty (TSA):
  All patients will receive a standard interscalene block with bupivacaine followed by indwelling catheter insertion with ropivacaine infusion to be left in place for two days.
  Interventions: Drug: Standard of care analgesia
- Liposomal bupivacaine (Experimental): THA:
  Standard of care analgesia, PLUS 266 mg of liposomal bupivacaine. Anterior capsule Inferior capsule Posterior capsule Short external rotator Gluteus maximus Subcutaneous tissue
  TKA:
  Standard of care analgesia, PLUS 266 mg of liposomal bupivacaine. Posterior knee capsule Anterior femoral periosteum Anterior tibial periosteum Subcutaneous tissue Pericapsular meniscal tissue
  TSA:
  All patients will receive a standard interscalene block with bupivacaine PLUS 266 mg of liposomal bupivacaine.
  Posterior capsule Rotator cuff Subscapularis Humeral periosteum Subcutaneous tissue Deltopectoral muscle
  Interventions: Drug: Liposomal bupivacaine; Drug: Standard of care analgesia

INTERVENTIONS:
Drug: Liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Standard of care analgesia
  Other Names: Bupivacaine; Ropivacaine; Fentanyl; Solumedrol; Morphine; Saline; Epinephrine

SUMMARY:
The purpose of this study is to determine whether liposomal bupivacaine is effective in the management of pain following total joint arthroplasty, as compared to standard of care analgesia.

DETAILED DESCRIPTION:
Liposomal bupivacaine (Exparel®) is a local anesthetic made up of liposomal encapsulated bupivacaine. It is designed to be injected at the time of surgery into the local soft tissues. Because of its unique liposomal delivery system, Liposomal bupivacaine (Exparel®) has been shown to provide up to 96 hours of pain relief following surgeries. This makes it an attractive option in total joint arthroplasty patients. Combined with the proven efficacy of regional anesthesia, intraoperative liposomal bupivacaine (Exparel®) may provide extended pain relief following total joint arthroplasty. This has the potential to avoid the need for opioid medications. With better pain control, medication side effects can be avoided and patient's length of stay in the hospital can be shortened.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of osteoarthritis
2. Elected to undergo primary TKA, THA, or TSA

Exclusion Criteria:

1. Age < 18 years
2. Pregnant or breastfeeding
3. Non-English speaking
4. Unable to give informed consent
5. Previous open hip, knee or shoulder surgery
6. Pre-determined patients discharging to ECF
7. Patients with allergies to bupivacaine
8. Patients currently taking opioid pain medication
9. Patients with contraindication to nerve blocks
10. Patients undergoing simultaneous bilateral joint replacement, as this would require >1 dose of liposomal bupivacaine (Exparel®) per patient for each surgical site
11. Patients with severe hepatic disease
12. Patients with chronic heart disease as defined as a decreased ejection fraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Napier, BSN,RN,MA, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth Riverside Methodist Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period July 1, 2014 to September 30, 2015 for patients undergoing total hip, knee or shoulder arthroplasty at OhioHealth Riverside Methodist Hospital.
Pre-assignment Details: Patients were randomized in a one to one fashion to one of two study groups within each surgical group. 10 patients were excluded after enrollment due to dual enrollment in another study, changes in anesthesia plan or improper dose of study drug. These 10 patients were not included in the analysis.
Groups:
- Standard of Care Analgesia: THA:
  33 patients received a spinal anesthetic using Fentanyl and Bupivacaine
  Injection into capsular tissue after placement of the acetabular component:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  TKA:
  39 patients received a spinal anesthetic using Fentanyl and Bupivacaine 39 patients received an adductor canal block of 0.25% Bupivacaine w/epinephrine 30cc
  Injection into posterior capsule of the knee:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  TSA:
  35 patients received a standard interscalene block with bupivacaine followed by indwelling catheter insertion with ropivacaine infusion to be left in place for two days.
  Standard of care analgesia
- Liposomal Bupivacaine: THA:
  36 patients received the standard of care analgesia, PLUS 266 mg of liposomal bupivacaine.
  Anterior capsule Inferior capsule Posterior capsule Short external rotator Gluteus maximus Subcutaneous tissue
  TKA:
  34 patients received the standard of care analgesia, PLUS 266 mg of liposomal bupivacaine.
  Posterior knee capsule Anterior femoral periosteum Anterior tibial periosteum Subcutaneous tissue Pericapsular meniscal tissue
  TSA:
  34 patient received a standard interscalene block with bupivacaine PLUS 266 mg of liposomal bupivacaine.
  Posterior capsule Rotator cuff Subscapularis Humeral periosteum Subcutaneous tissue Deltopectoral muscle
  Liposomal bupivacaine
  Standard of care analgesia
Period: Overall Study
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine
Started | 107 | 104
Completed | 107 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Analgesia: THA:
  All patients will receive a spinal anesthetic using Fentanyl and Bupivacaine
  Injection into capsular tissue after placement of the acetabular component:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  TKA:
  All patients will receive a spinal anesthetic using Fentanyl and Bupivacaine All patients will receive an adductor canal block of 0.25% Bupivacaine w/epinephrine 30cc
  Injection into posterior capsule of the knee:
  0.5% Bupivacaine 15 cc 40 mg Solumedrol 10 mg Morphine 20 cc Saline
  TSA:
  All patients will receive a standard interscalene block with bupivacaine followed by indwelling catheter insertion with ropivacaine infusion to be left in place for two days.
  Standard of care analgesia
- Liposomal Bupivacaine: THA:
  Standard of care analgesia, PLUS 266 mg of liposomal bupivacaine. Anterior capsule Inferior capsule Posterior capsule Short external rotator Gluteus maximus Subcutaneous tissue
  TKA:
  Standard of care analgesia, PLUS 266 mg of liposomal bupivacaine. Posterior knee capsule Anterior femoral periosteum Anterior tibial periosteum Subcutaneous tissue Pericapsular meniscal tissue
  TSA:
  All patients will receive a standard interscalene block with bupivacaine PLUS 266 mg of liposomal bupivacaine.
  Posterior capsule Rotator cuff Subscapularis Humeral periosteum Subcutaneous tissue Deltopectoral muscle
  Liposomal bupivacaine
  Standard of care analgesia
- Total: Total of all reporting groups
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 107 | 104 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.4) | 65.9 (9.1) | 66.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 61 | 118
  Male | 50 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in Hospital (Days)
Time Frame: Participants were followed for the duration of hospital stay, an expected average of 3 days
Measure: Median (Full Range); unit: days
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine
Number analyzed (Participants) | 107 | 104
days | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 3.0]
Statistical Analysis 1: Comparison: Standard of Care Analgesia vs Liposomal Bupivacaine; Test type: Superiority or Other; p = 0.764, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to Post-operative Rescue Opioids (Hours)
Time Frame: Immediately following discharge from operating room until the participant was discharged from the hospital, an expected average of 3 days
Measure: Median (Full Range); unit: hours
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine
Number analyzed (Participants) | 107 | 104
hours | 7.7 [2.6 to 49.5] | 11.8 [2.2 to 75.0]
Statistical Analysis 1: Comparison: Standard of Care Analgesia vs Liposomal Bupivacaine; Test type: Superiority or Other; p = 0.206, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Readmission or Emergency Department (ED) Visit Due to Pain Control Within 30 Days
Time Frame: Date of discharge through 30 days following discharge
Measure: Number; unit: participants
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine
Number analyzed (Participants) | 107 | 104
participants | 2 | 4
Statistical Analysis 1: Comparison: Standard of Care Analgesia vs Liposomal Bupivacaine; Test type: Superiority or Other; p = 0.656, Fisher Exact; Fisher exact = 0.486

ADVERSE EVENTS:
Groups:
- Liposomal Bupivacaine: THA:
  36 patients received the standard of care analgesia, PLUS 266 mg of liposomal bupivacaine.
  Anterior capsule Inferior capsule Posterior capsule Short external rotator Gluteus maximus Subcutaneous tissue
  TKA:
  33 patients received the standard of care analgesia, PLUS 266 mg of liposomal bupivacaine.
  Posterior knee capsule Anterior femoral periosteum Anterior tibial periosteum Subcutaneous tissue Pericapsular meniscal tissue
  TSA:
  34 patient received a standard interscalene block with bupivacaine PLUS 266 mg of liposomal bupivacaine.
  Posterior capsule Rotator cuff Subscapularis Humeral periosteum Subcutaneous tissue Deltopectoral muscle
  Liposomal bupivacaine
  Standard of care analgesia
Arm/Group | Standard of Care Analgesia | Liposomal Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/104
Other Adverse Events (participants affected / at risk) | 0/107 | 2/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Analgesia (N=107) | Liposomal Bupivacaine (N=104)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
No early termination or technical problems identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No